CLINICAL TRIAL: NCT06911788
Title: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD, SINGLE-DOSE, CROSS-OVER STUDY TO ESTIMATE THE ABSOLUTE BIOAVAILABILITY OF VEPDEGESTRANT (ARV-471, PF-07850327) FOLLOWING ORAL AND INTRAVENOUS DOSING OF THE DRUG TO HEALTHY PARTICIPANTS
Brief Title: A Study to Learn How a Tablet Compared With an IV Infusion of the Study Medicine Called Vepdegestrant is Taken up Into the Blood in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4891037; 2024-518134-92-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vepdegestrant oral and IV administration (Experimental): Participants will receive a single IV infusion of Vepdegestrant on Day 1 of Period 1 followed by a single 200 mg dose of Vepdegestrant registrational tablet on Day 1 of Period 2.
  Interventions: Drug: Vepdegestrant (Reference); Drug: Vepdegestrant (Test)

INTERVENTIONS:
Drug: Vepdegestrant (Reference) — Participants will receive a single intravenous (IV) dose of Vepdegestrant on Period 1 Day 1
  Other Names: ARV-471, PF-07850327
Drug: Vepdegestrant (Test) — Participants will receive a 200 mg single oral dose of Vepdegestrant tablet formulation on Period 2 Day 1
  Other Names: ARV-471, PF-07850327

SUMMARY:
The purpose of this study is to learn how much of the study medicine called Vepdegestrant will reach the bloodstream when given orally compared to given intravenously.

This study is seeking participants who:

* are healthy males and healthy females who cannot have children.
* are 18 years or older.
* are healthy as decided by medical tests.
* have a body mass index (BMI) of 16 to 32 kilogram per meter squared.
* have a total body weight of more than 45 kilograms (99 pounds).

In Period 1, all participants will receive one dose of Vepdegestrant by IV. In Period 2, all participants will receive one dose of Vepdegestrant by mouth following a high-fat breakfast. The levels of Vepdegestrant in Period 1 will be compared to the levels of Vepdegestrant in Period 2 and the bioavailablility of the oral formulation of Vepdegestrant will be determined.

The study duration is 22 days and includes two periods. Participants will stay in the clinical research unit for 9 days (8 nights) during each period. A follow-up visit for each participant takes place at 28 to 35 days after taking the study medicine for the last time.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male participants, and/or female participants of non-childbearing potential who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
2. Body mass index (BMI) of 16-32 kg/m2; and a total body weight >45 kg (99 lb).

Key Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy)
   * History of or positive testing for HIV infection, hepatitis B, or hepatitis C.
2. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements, grapefruit/grapefruit containing products, and Seville orange/Seville orange containing products within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
4. Previous administration with an investigational product (drug or vaccine) within 30 days or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
5. A positive urine drug test
6. Screening blood pressure ≥140/90 mm Hg for participants <60 years; and ≥150/90 mm Hg for participants ≥60 years old.
7. Renal impairment as defined by an eGFR in adults <60 mL/min/1.73 m² based on CKD-EPI equation.
8. Standard 12 lead electrocardiogram that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete left bundle branch block, signs of a myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias).
9. History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
10. 6 months prior or current use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.
11. History of sensitivity to heparin or heparin-induced thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Dose-normalized (dn) Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Vepdegestrant after oral administration | At predefined intervals throughout the treatment period, up to approximately 1 week after the last dose of Vepdegestrant
  dn AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞) divided by dose. It is obtained from AUC (0 - t) plus AUC (t - ∞).
Dose-normalized (dn) Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Vepdegestrant after IV administration | At predefined intervals throughout the treatment period, up to approximately 1 week after the last dose of Vepdegestrant
  dn AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | First dose of Vepdegestrant through 35 days after last dose Vepdegestrant
Number of Participants With Clinical Laboratory Abnormalities | First dose of Vepdegestrant through 35 days after last dose Vepdegestrant
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | First dose of Vepdegestrant through 35 days after last dose Vepdegestrant
Number of Participants With Electrocardiogram (ECG) Abnormalities | First dose of Vepdegestrant through 35 days after last dose Vepdegestrant

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Netherlands (2):
  - ICON, Groningen
  - ICON - screening centre, Utrecht

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891037